CLINICAL TRIAL: NCT06840535
Title: A Phase I Study to Evaluate the Safety and Dosimetry of 68Ga-OncoACP3 in Patients With Prostate Cancer
Brief Title: A Study to Evaluate the Safety and Dosimetry of 68Ga-OncoACP3 in Patients With Prostate Cancer
Acronym: OncoACP-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PH-ACP3GA-01/24; 2024-515608-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic Disease; PSA Level Greater Than 0.2
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are divided into two cohorts:
  * Cohort A: 5 male patients without visceral or bone metastases, which would interfere with dosimetry evaluation of healthy organs.
  * Cohort B: all patients who meet the eligibility criteria (up to 15 patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coort A (Experimental): 5 male patients without visceral or bone metastases, which would interfere with dosimetry evaluation of healthy organs.
- Coort B (Experimental): All patients who meet the eligibility criteria (up to 15 patients)
  Interventions: Drug: [68Ga]Ga-OncoACP3

INTERVENTIONS:
Drug: [68Ga]Ga-OncoACP3 — Single intravenous bolus injection.
  Arms: Coort B

SUMMARY:
The aim of this study is to assess the safety and dosimetry of [68Ga]Ga-OncoACP3 in patients with prostate cancer.

DETAILED DESCRIPTION:
The Acid Phosphatase 3 (ACP3) is expressed in primary and metastatic prostate cancer lesions. OncoACP3 is a new ligand for ACP3.

This is a phase I, multicenter clinical trial to evaluate the safety, dosimetry and biodistribution of [68Ga]Ga-OncoACP3 as a PET radiotracer for the diagnostic imaging of prostate cancer. In this trial, 68Ga-OncoACP3 is offered to prostate cancer patients who already received standard of care imaging and might therefore complement available modalities.

Eligible patients for this trial are prostate cancer patients, aged 18 years or more with:

* suspected metastasis who are candidates for initial definitive therapy
* suspected recurrence based on elevated serum prostate-specific antigen (PSA) level (i.e., a progressive and confirmed serum PSA level > 0.2 ng/mL)
* metastatic disease who might be candidates for treatment with 177Lu-labelled PSMA ligands

All patients will undergo PET/CT imaging with [68Ga]Ga-OncoACP3.

Patients are divided into two cohorts:

* Cohort A: 5 male patients without visceral or bone metastases, which would interfere with dosimetry evaluation of healthy organs.
* Cohort B: all patients who meet the eligibility criteria (up to 15 patients)

Both cohorts are recruited in parallel, and patients are assigned to the respective cohort based on their disease extent. Whenever possible, patients are enrolled in cohort A, unless they are unsuitable for cohort A, or the required number of patients has already been enrolled in cohort A.

All patients will receive a single intravenous bolus administration of [68Ga]Ga-OncoACP3 and biodistribution, PK, and dosimetry of [68Ga]Ga-OncoACP3 will be assessed based on a series of PET/CT scans, blood and urine sampling.

Full dosimetry evaluations will be performed for all patients in cohort A. Dosimetry in the other patients may be performed to the extent that it is possible based on their disease burden (i.e., only organs not affected by malignant lesions can be evaluated), as appropriate.

All patients will be assessed for safety. In addition, relative uptake to appropriate reference tissue of [68Ga]Ga-OncoACP3 as well as semiquantitative parameters such as SUVmax/SUVmean/SUVsd, are determined. The correlation of [68Ga]Ga-OncoACP3 uptake with immunopathology staining for ACP3 will be evaluated in patients undergoing surgery or tumor biopsy collection. For patients who undergo PSMA-PET/CT within 4 weeks before or after the [68Ga]Ga-OncoACP3-PET/CT scan, the lesion detection rate will be compared Full dosimetry evaluations will be performed for all patients in cohort A. Additional dosimetry in the other patients may be performed to the extent that it is possible based on their disease burden (i.e., only organs not affected by malignant lesions can be evaluated).

ELIGIBILITY:
Inclusion Criteria:

1. Prostate cancer patients with:

   * suspected metastasis who are candidates for initial definitive therapy
   * suspected recurrence based on elevated serum prostate-specific antigen (PSA) level (i.e., a progressive and confirmed serum PSA level > 0.2 ng/mL)
   * metastatic disease who might be candidates for treatment with 177Lu-labelled PSMA ligands
2. Patients with a negative PSMA-PET/CT or discordant PSMA PET and FDG-PET findings are eligible for this study, providing that they have a confirmed diagnosis of prostate cancer.
3. Subjects able to father children must agree to practice effective contraception for three months starting from the study drug administration.
4. Age ≥ 18
5. ECOG ≤ 1
6. Patient must not have any concomitant infections or active concomitant disease.
7. All acute toxic effects (excluding alopecia and fatigue) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v. 5.0) Grade ≤ 1.
8. Life expectancy of more than 12 weeks.
9. Ability to undergo imaging study procedures.
10. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
11. Willingness and ability to comply with the scheduled visits, plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Chronically impaired renal function as expressed by creatinine clearance < 60 mL/min or serum creatinine > 1.5 x ULN.
2. Presence of active hepatitis.
3. Presence of significant cardiac disorders (congestive heart failure, NYHA class III-IV, myocardial infarction within one year prior to study entry, uncontrolled hypertension, or arrhythmia).
4. Any concomitant condition which in the opinion of investigators makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
5. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of the study drug. Minimally invasive procedures such as biopsies are not considered as exclusion criteria.
6. Serious, non-healing wound, ulcer, or bone fracture.
7. Allergy to study medication or excipients in study medication.
8. Any anti-cancer therapy (e.g., cytotoxic chemotherapy, immunotherapy, radiation, surgery, etc.) within 3 weeks before [68Ga]Ga-OncoACP3-PET/CT scan.
9. Subject has received, or is scheduled to receive, another investigational medicinal product (IMP) from one month before [68Ga]Ga-OncoACP3 injection to end of study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Cohort A: Dosimetry - Effective dose equivalent (mSv) | Assessed on day 1
  Whole-body effective dose (mSv) following administration of a single dose of [68Ga]Ga-OncoACP3.
Cohort A: Dosimetry - Effective dose absorbed doses (mGy) | Assessed on day 1
  Absorbed doses (mGy) of normal organs following administration of a single dose of [68Ga]Ga-OncoACP3.
All patients: Safety (AEs and SAEs) | Throughout study, until a maximum of 7 days after the administration of the study drug.
  Safety of administration of [68Ga]Ga-OncoACP3, assessed based on Common Toxicity Criteria (CTCAE version 5.0)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) - Blood | Assessed on day 1
  Pharmacokinetics (PK) of [68Ga]Ga-OncoACP3 based on measurement on blood of residual radioactivity over time [kBq/mL]
Excretion - Urine | Assessed on day 1
  Excretion of [68Ga]Ga-OncoACP3 based on measurement of residual radioactivity in the urine over time [kBq]
Biodistribution profile: SUVmax | Assessed on day 1
  Uptake of [68Ga]Ga-OncoACP3 in tumor lesions and healthy organs in terms of SUVmax
Biodistribution profile: SUVmean | Assessed on day 1
  Uptake of [68Ga]Ga-OncoACP3 in tumor lesions and healthy organs in terms of SUVmean
Biodistribution profile: SUVsd | Assessed on day 1
  Uptake of [68Ga]Ga-OncoACP3 in tumor lesions and healthy organs in terms of SUVsd

OTHER OUTCOMES:
Immunopathology staining | Within 8 weeks of the scan, surgery and biopsy collection
  Correlation of the uptake of [68Ga]Ga-OncoACP3 with immunopathology staining for ACP3 expression and comparison to staining for PSMA expression, in all patients for whom surgical or biopsy specimen are available.
Lesion detection rate | The [68Ga]Ga-OncoACP3-PET/CT scan needs to be collected within 4 weeks
  Lesion detection rate compared to PSMA-PET/CT.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - ASST Papa Giovanni XXIII, Bergamo, BG
  - IRCCS Ospedale San Raffaele, Milan, Milano
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milano

IPD SHARING:
Plan to Share IPD: No